CLINICAL TRIAL: NCT01113541
Title: A One-year, Phase III, Open-label, Non-comparative Trial of the Effect of Ziprasidone HCl on Metabolic Syndrome Risk Factors in Patients With Bipolar Disorder
Brief Title: One-Year Trial of Oral Ziprasidone in Bipolar Patients With Metabolic Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281190
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Bipolar Disorder
Keywords: Ziprasidone; Bipolar Disorder; Metabolic Syndrome
MeSH Terms: conditions — Bipolar Disorder; Metabolic Syndrome | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active treatment (switch to oral Ziprasidone) (Experimental)
  Interventions: Drug: Ziprasidone HCL (oral)

INTERVENTIONS:
Drug: Ziprasidone HCL (oral) — Ziprasidone Hydrochloride 20 to 80 mg administered orally twice a day (40-160 mg total daily dose) for up to 1 year.
  Other Names: Zeldox, Geodon

SUMMARY:
The purpose of this study is to explore the impact of Ziprasidone HCl on the distribution of metabolic syndrome (MS) risk factors in a population of Bipolar patients presenting with glucose intolerance, dyslipidemia and/or elevated waist circumference associated with their current antipsychotic medication.

DETAILED DESCRIPTION:
The trial was terminated prematurely on December 14, 2010, due to inability to recruit the planned number of subjects and shifting organizational priorities. The decision to terminate the trial was not based on any safety or efficacy concerns.

ELIGIBILITY:
Inclusion Criteria:

* Subject must present at least 2 of the following risk factors of MS at screening: Elevated waist circumference: >102 cm in men and >88 cm in women; Elevated triglycerides (TGs): ≥1.7 mmol/L (≥150 mg/dL); Reduced HDL-Cholesterol: <1.03 mmol/L (<40 mg/dL) in men and <1.3 mmol/L (<50 mg/dL) in women; Elevated fasting glucose: ≥ 5.6 mmol/L.
* According to the clinical judgment of the investigator, the risk factors for MS have developed in close temporal relationship to starting an antipsychotic medication.
* Substitution to a less metabolically disruptive antipsychotic medication is considered

Exclusion Criteria:

* Subjects with contraindication(s) to the use of Ziprasidone according to Canadian prescribing information.
* Subjects with a history of treatment resistance.
* Subjects with any medical condition (e.g. pre-existing diabetes, pre-existing dyslipidemia, thyroid pathology) or taking any concomitant medication (e.g. topiramate or other weight loss-promoting agents, hypoglycemic agents, hypolipemic agents), that may confound the evaluation of the study drug.
* Body mass index ≥ 40 at baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Canada (10):
  - Foothills Medical Centre, Department of Psychiatry, Calgary, Alberta
  - Mental Health Centre for Research and Education, Calgary, Alberta
  - Dr. Alexander McIntyre Inc., Penticton, British Columbia
  - Country Club Plaza, Winnipeg, Manitoba
  - Edgeland Medical, Dr. Alla Kirshner Medical Corporation, Winnipeg, Manitoba
  - Capital, Health Authority, QE II Health Sciences Centre, Mood Disorder Clinic, Halifax, Nova Scotia
  - Office of Dr. A. K. Munshi, Sydney, Nova Scotia
  - Centre de recherche Fernand-Seguin de l'hopital Louis H. Lafontaine, Montreal, Quebec
  - Clinique St-Leonard, Montreal, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281190&StudyName=One-Year%20Trial%20of%20Oral%20Ziprasidone%20in%20Bipolar%20Patients%20with%20Metabolic%20Syndrome%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-seven participants were screened for the study and 13 participants were assigned to study drug and treated.
Groups:
- Ziprasidone: Days 1 to 3: 40 milligrams (mg) twice daily (BID); Days 4 to 7: 60 mg BID; Days 8 to15: 80 mg BID; Day 16 to Week 52: 20-80 mg BID flexible dosing.
Period: Overall Study
Arm/Group | Ziprasidone
Started | 13
Completed | 0
Not Completed | 13
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Not completed — Study Terminated by Sponsor | 7
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Ziprasidone
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Reduction From Baseline of at Least 1 Risk Factor for Metabolic Syndrome (MS) at Week 52 or Premature Discontinuation
Description: MS risks factors: elevated (el) waist circumference: ≥102 centimeters (cm) in men and ≥88 cm in women (Asian origin: ≥90 cm [men] and ≥80 cm [women]); el triglycerides: ≥1.7 millimoles per liter (mmol/L) (1≥50 milligrams per deciliter [mg/dL]); reduced high-density lipoprotein cholesterol (HDL-C): <1.03 mmol/L (<40 mg/dL) in men and <1.3 mmol/L (<50 mg/dL) in women; el fasting glucose: ≥5.6 mmol/L (≥100 mg/dL); and el systolic/diastolic blood pressure: systolic ≥130 millimeters of mercury (mmHg) and/or diastolic ≥85 mmHg. Responder = at least 1 less risk factor at endpoint than baseline.
Time Frame: Week 52 or Early Termination
Population: Per protocol population: all subjects in the intent-to-treat population who remained in the study for at least 28 weeks. N = number of participants with analyzable data at observation.
Measure: Number; unit: percentage of participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 10
percentage of participants | 50.00

2. Secondary Outcome: Mean Change From Baseline in the Number of Risk Factors of Metabolic Syndrome (MS)
Description: MS risks factors: elevated waist circumference: ≥102 cm in men and ≥88 cm in women (Asian origin: ≥90 cm [men] and ≥80 cm [women]); elevated triglycerides: ≥1.7 mmol/L (1≥50 mg/dL); reduced HDL-C: <1.03 mmol/L (<40 mg/dL) in men and <1.3 mmol/L (<50 mg/dL) in women; elevated fasting glucose: ≥5.6 mmol/L (≥100 mg/dL); and elevated systolic/diastolic blood pressure: systolic blood pressure ≥130 mm Hg and/or diastolic blood pressure ≥85 mm Hg.
Time Frame: Baseline, Week 52
Population: PP and Intent-to-treat (ITT) population; ITT population = all participants enrolled in the study who received at least 1 dose of study medication and who had baseline and at least 1 post-baseline MS measurement. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

3. Secondary Outcome: Metabolic Syndrome (MS) Prevalence
Description: Percentage of participants at each visit defined as having metabolic syndrome (MS) based on the National Cholesterol Education Program (NCEP) Adult Treatment Panel III. MS = 3 or more of 5 characteristics: abdominal obesity, hypertriglyceridemia, low high-density lipoprotein (HDL) cholesterol, high blood pressure, and high fasting glucose.
Time Frame: Baseline through Week 52
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in the Percentage of Participants With Each Individual Metabolic Syndrome (MS) Risk Factor
Description: as for outcome 2
Time Frame: Baseline through Week 52
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

5. Secondary Outcome: Percentage of Participants With Individual Metabolic Syndrome (MS) Risk Factors
Description: MS risks factors = elevated waist circumference: ≥102 cm in men and ≥88 cm in women (Asian origin: ≥90 cm [men] and ≥80 cm [women]); elevated triglycerides: ≥1.7 mmol/L (1≥50 mg/dL); reduced HDL-C: <1.03 mmol/L (<40 mg/dL) in men and <1.3 mmol/L (<50 mg/dL) in women; elevated fasting glucose: ≥5.6 mmol/L (≥100 mg/dL); and elevated systolic/diastolic blood pressure: systolic blood pressure ≥130 mm Hg and/or diastolic blood pressure ≥85 mm Hg.
Time Frame: Baseline through Week 52
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Individual Risk Factors of Metabolic Syndrome (MS): Elevated Waist Circumference
Description: MS risk factor elevated waist circumference defined as ≥102 centimeters (cm) in men and ≥88 cm in women (Asian origin: ≥90 cm [men] and ≥80 cm [women]).
Time Frame: Baseline, Week 4, Week 12, Week 52
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline in Individual Risk Factors of Metabolic Syndrome (MS): Elevated Systolic/Diastolic Blood Pressure
Description: MS risk factor elevated systolic/diastolic blood pressure defined as systolic blood pressure ≥130 millimeters of mercury (mm Hg) and/or diastolic blood pressure ≥85 mm Hg.
Time Frame: Baseline, Week 4, Week 12, Week 52
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Individual Risk Factors of Metabolic Syndrome (MS): Elevated Fasting Glucose
Description: MS risk factor elevated fasting glucose defined as ≥5.6 millimoles per liter (mmol/L) (≥100 mg/dL).
Time Frame: Baseline, Week 4, Week 12, Week 52
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

9. Secondary Outcome: Change From Baseline in Individual Risk Factors of Metabolic Syndrome (MS): Reduced High-density Lipoprotein Cholesterol (HDL-C)
Description: MS risk factor reduced HDL-C defined as <1.03 millimoles per liter (mmol/L) (<40 mg/dL) in men and <1.3 mmol/L (<50 mg/dL) in women.
Time Frame: Baseline, Week 4, Week 12, Week 52
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline in Individual Risk Factors of Metabolic Syndrome (MS): Elevated Triglycerides
Description: MS risk factor elevated triglycerides defined as ≥1.7 millimoles per liter (mmol/L) (1≥50 mg/dL).
Time Frame: Baseline, Week 4, Week 12, Week 52
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

11. Secondary Outcome: Change From Baseline in Ten-year Coronary Heart Disease (CHD) Risk According to Framingham Scoring System
Description: Framingham scoring system risk factors: age (risk points range: -9 to 16), cholesterol (risk points range: 0 to 13), HDL cholesterol (risk points range: -1 to 2), smoking (risk points range: 0 to 9), and systolic blood pressure (risk points range: 0 to 6); total risk points range <0 to ≥25, higher score indicates higher 10 year risk (range <1% to ≥30% 10 year risk).
Time Frame: Baseline, Week 4, Week 52
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

12. Secondary Outcome: Change From Baseline in Total Cholesterol and Low-density Lipoprotein (LDL) Cholesterol Levels
Time Frame: Baseline, Week 52 or Early Termination
Population: PP and ITT. Median was reported due to small sample size and risk of skewing.
Measure: Median (Full Range); unit: milligrams per deciliter
Arm/Group | Ziprasidone
Number analyzed (Participants) | 10
milligrams per deciliter
  Total cholesterol: Baseline | 206.0 [138.610 to 269.884]
  Total cholesterol: Change at Last Observation | -20.0 [-47.104 to 18.919]
  LDL cholesterol: Baseline | 131.0 [78.764 to 167.567]
  LDL cholesterol: Change at Last Observation | -8.0 [-36.680 to 16.988]

13. Secondary Outcome: Change From Baseline in Weight
Time Frame: Baseline, Week 4, Week 12, Week 52 or Early Termination
Population: PP and ITT; n = number of participants with evaluable data at observation.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Ziprasidone
Number analyzed (Participants) | 13
kilograms
  Baseline (n=13) | 93.5 (23.12)
  Value at Week 4 (n=9) | 92.9 (21.99)
  Value at Week 12 (n=5) | 97.3 (25.37)
  Value at Week 52 (n=10) | 87.5 (24.50)

14. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Body mass index = weight in kilograms (kg) / height in meters (m)^2 .
Time Frame: Baseline, Week 4, Week 12, Week 52 or Early Termination
Population: PP and ITT. Results for BMI not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

15. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Time Frame: Baseline, Week 52 or Early Termination
Population: PP and ITT. Median was reported due to small sample size and risk of skewing. Last observation = last observation while on study drug or during the lag.
Measure: Median (Full Range); unit: percent HbA1c
Arm/Group | Ziprasidone
Number analyzed (Participants) | 10
percent HbA1c
  Baseline | 5.5 [5.3 to 6.1]
  Median change | -0.2 [-0.3 to 0.1]

16. Secondary Outcome: Change From Baseline in Insulin Levels
Time Frame: Baseline, Week 52 or Early Termination
Population: PP and ITT. Insulin levels not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

17. Secondary Outcome: Change From Baseline in Corrected QT Interval (QTc): Fridericia's Heart Rate Correction Formula (QTcF)
Description: QT interval is the time between the start of the Q wave and the end of the T wave in the cardiac electrical cycle. QTc is the QT interval corrected for heart rate. Corrected QT interval using Fridericia's heart rate correction formula: QTcF = QT/RR^1/3, where RR=RR interval in seconds.
Time Frame: Baseline, Week 4, Week 52 or Early Termination
Population: PP and ITT; n = number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Ziprasidone
Number analyzed (Participants) | 13
milliseconds
  Baseline (n=13) | 421.0 (12.16)
  Week 4 (n=9) | 434.0 (13.61)
  Week 52 or or Early Termination (n=9) | 428.8 (14.65)

18. Secondary Outcome: Change From Baseline in Apolipoprotein B (ApoB) Levels
Time Frame: Baseline, Week 52 or Early Termination
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

19. Secondary Outcome: Change From Baseline in Leptin
Time Frame: Baseline, Week 52 or Early Termination
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

20. Secondary Outcome: Change From Baseline in Physical Activity Index
Description: Physical activity (exercise) score derived for each participant based on the frequency and intensity of physical activities: regular walking, recreational activity, cycling, and sporting activity. Six categories of total score: inactive (range: 0-2), occasional (range: 3-5), light (range: 6-8), moderate (range: 9-12), moderately vigorous (range: 13-20), and vigorous (≥21). Higher score = higher frequency and intensity of physical activity.
Time Frame: Baseline, Week 28, Week 52 or Early Termination
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

21. Secondary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) - Total Score
Description: Measures the overall severity of depressive symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Baseline, Week 4, Week 12, Week 28, Week 52 or Early Termination
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

22. Secondary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS)
Description: 11-item scale that measures the severity of manic episodes from subject reported symptoms over previous 48 hours and clinical observation during interview. Four items (irritability, speech, thought content, disruptive-aggressive behaviour) are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining 7 items (elevated mood, increased motor activity-energy, sexual interest, sleep, language-thought disorder, appearance, insight) are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). YMRS total score range = 0 to 60.
Time Frame: Baseline, Week 4, Week 12, Week 28, Week 52 or Early Termination
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

23. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Subscale
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected.
Time Frame: Baseline, Week 4, Week 12, Week 28, Week 52 or Early Termination
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

24. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Subscale Score
Description: CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Week 52 or Early Termination
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

25. Secondary Outcome: Change From Baseline in Drug Attitude Inventory (DAI)
Description: DAI, a 10-item scale to assess how the attitude of schizophrenia participants toward their medications may affect compliance. Respondents indicate 'true' or 'false' for each item. An overall calculated score ranged from -10 to 10, where a positive score indicated a positive subjective response (compliant), a negative score indicated non-compliance. Change: score at observation minus score at baseline.
Time Frame: Week 28, Week 52 or Early Termination
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

26. Secondary Outcome: Change From Baseline in Social and Occupational Functioning Assessment Scale (SOFAS)
Description: 0-100 single score scale focusing exclusively on participant's level of social and occupational functioning; not directly influenced by overall severity of participant's psychological symptoms; higher score = higher level of functioning. 1 to 10 = persistent inability to maintain minimal personal hygiene; unable to function without harming self or others or without considerable external support; 91 to 100 = superior functioning in a wide range of activities.
Time Frame: Baseline, Week 28, Week 52 or Early Termination
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

27. Secondary Outcome: Change From Baseline in EuroQoL Index (EQ-I)
Description: EQ-5D: subject rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (confined to bed). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Week 28, Week 52 or Early Termination
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

28. Secondary Outcome: Change From Baseline in European Quality of Life (EuroQol) Visual Analogue Scale (EQ-5D VAS): Current Health State Score
Description: EQ-5D: subject rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline, Week 28, Week 52 or Early Termination
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

29. Secondary Outcome: Change From Baseline in Impact of Weight on Quality of Life-Lite Version (IWQOL-Lite) Scale
Description: 31-item self report inventory to assess impact of weight on quality of life. Five subscales: physical functioning, self-esteem, sexual life, public distress, and work, with categories in each subscale scored 1 (no trouble or difficulty) to 5 (persistent trouble or difficulty). The rescaled IWQoL-Lite score is determined by the sum of scores on all 31 items and rescaling this sum to a 1 to 100 scoring with 0=the poorest and 100=the best quality of life.
Time Frame: Baseline, Week 28, Week 52 or Early Termination
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

30. Secondary Outcome: Number of Participants With Suicidal Tendencies (Columbian-Suicide Severity Rating Scale, [C-SSRS], Mapped to C-CASA [Columbia Classification Algorithm For Suicide Assessment])
Description: C-SSRS is a participant rated questionnaire to assess suicidal ideation, suicidal behavior, actual attempts (yes or no responses), and intensity of ideation (rated 1=low severity to 5=high severity). Yes/No responses are mapped to Columbia Classification Algorithm of Suicide Assessment (C-CASA) categories: Completed suicide, suicide attempt, preparatory acts toward imminent suicidal behavior, suicidal ideation, and self-injurious behavior, or no suicidal intent. A participant could have a yes or no response in more than one category.
Time Frame: Baseline, Week 1 through Week 52 or Early Termination
Population: PP and ITT. Results not reported: data not summarized due to limited enrollment and early termination of the study.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Ziprasidone
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=13)
Akathisia (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=13)
Vertigo (Ear and labyrinth disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Non-cardiac chest pain (General disorders) | 1
Thirst (General disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Blood cholesterol increased (Investigations) | 1
Blood prolactin increased (Investigations) | 1
High density lipoprotein decreased (Investigations) | 1
Low density lipoprotein increased (Investigations) | 1
Protein urine present (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Akathisia (Nervous system disorders) | 3
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 5
Memory impairment (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 4
Tension headache (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Emotional disorder (Psychiatric disorders) | 1
Flat affect (Psychiatric disorders) | 1
Hypomania (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 6
Mania (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Terminal insomnia (Psychiatric disorders) | 1
Menstruation irregular (Reproductive system and breast disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
This study was terminated due to slow enrollment and changes in organizational strategy and resources; most of the planned analyses in the statistical analysis plan were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.